CLINICAL TRIAL: NCT06018623
Title: Lean Body Weight Scalar for the Anesthetic Induction Dose of Propofol
Brief Title: Dosage of Propofol Based on Lean Body Weight
Status: Not yet recruiting | Type: Observational
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, DUYGU DEMİROZ, dr, Inonu University
Other Study IDs: TOTM
Record Dates: First submitted 2023-08-09; First posted 2023-08-30 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Gender; Anesthesia
Keywords: the lean body weight, propofol intubation conditions
MeSH Terms: conditions — Coitus

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- grup 1.Optimum range: Group 1 BMI = 18.5-24.9,
  Interventions: Other: It is an observational study and no non-routine procedures will be performed on patients. Routine anesthesia procedure will be applied to the patients
- Group 2.Overweight: BMI = 25-29.9,
  Interventions: Other: It is an observational study and no non-routine procedures will be performed on patients. Routine anesthesia procedure will be applied to the patients
- Group 3.Class I obesity: BMI=30-34.9
  Interventions: Other: It is an observational study and no non-routine procedures will be performed on patients. Routine anesthesia procedure will be applied to the patients

INTERVENTIONS:
Other: It is an observational study and no non-routine procedures will be performed on patients. Routine anesthesia procedure will be applied to the patients — It is an observational study and no non-routine procedures will be performed on patients.
  Routine anesthesia procedure will be applied to the patients

SUMMARY:
Patients who will be anesthesia induced with propofol will be body analyzed with Tanita before the operation. Height, weight, age, gender and other general information of the patients will be recorded. Total body weight (TBW), ideal body weight (IBW) and lean body weight (LBW) will be calculated. Patients over 18 years of age who will be operated under general anesthesia for 2-6 hours will be included. Patients allergic to propofol or contraindicated to propofol will be excluded. In the study, in order to decide and test the most appropriate weight-based scale for the evaluation of propofol dosage for induction of anesthesia by identifying patients who need additional propofol during intubation, Ingrande et al. After monitoring, propofol infusion (100 mg/kg/hour) will be started according to total body weight and the infusion will be stopped when the BIS value is between 50 and 40 and the elapsed time will be recorded. Routine anesthesia applications will be performed by applying neuromuscular blocker. Total Propofol dose administered will be calculated according to the dose TBW, IBW and LBW in kilograms. The relationship between the doses administered and body mass index will be evaluated.

DETAILED DESCRIPTION:
Patients who will be anesthesia induced with propofol will be body analyzed with Tanita before the operation. Height, weight, age, gender and other general information of the patients will be recorded. Total body weight (TBW), ideal body weight (IBW) and lean body weight (LBW) will be calculated. Patients over 18 years of age who will be operated under general anesthesia for 2-6 hours will be included. Patients who are allergic to propofol or for whom propofol is contraindicated will not be included in the study. In the study, 80 patients with a mean body mass index [BMI] between 18-35 and Bispectoral index (BIS) (Ingrande et al. ) monitoring, propofol infusion (100 mg/kg/hour) will be started according to total body weight, and when the BIS value is between 50 and 40, the infusion will be stopped and the elapsed time will be recorded in order to decide and test the most appropriate weight-based scale for propofol dosing for anesthesia induction to identify and evaluate patients who need additional propofol during intubation. Routine anesthesia will be performed by applying neuromuscular blocker. Total Propofol dose administered will be calculated according to TBW, IBW and LBW per kilogram. And the relationship between the doses given and body mass index will be evaluated. In our study, we aimed to evaluate the effects of Propofol dose according to lean body weight by evaluating patients with a body mass index below 35.Patients who will undergo anesthesia induction with Propofol will undergo preoperative body analysis with Tanita. Height, weight, age, gender and other general information of the patients will be recorded. Total body weight (TBW), ideal body weight (IBW) and lean body weight (LBW) will be calculated. Patients over 18 years of age who will be operated under general anesthesia for 2-6 hours will be included. Patients who are allergic to propofol or for whom propofol is contraindicated will not be included in the study. In the study, 80 patients with a mean body mass index [BMI] between 18-35 and Bispectoral index (BIS) (Ingrande et al. ) monitoring, propofol infusion (100 mg/kg/hour) will be started according to total body weight, and when the BIS value is between 50 and 40, the infusion will be stopped and the elapsed time will be recorded in order to decide and test the most appropriate weight-based scale for propofol dosing for anesthesia induction to identify and evaluate patients who need additional propofol during intubation. Routine anesthesia will be performed by applying neuromuscular blocker. Total Propofol dose administered will be calculated according to TBW, IBW and LBW per kilogram. And the relationship between the doses given and body mass index will be evaluated. In our study, we aimed to evaluate the effects of Propofol dose according to lean body weight by evaluating patients with a body mass index below 35.

ELIGIBILITY:
Inclusion Criteria: BMI 18-35 will be included. over 18 years old It will take 2-6 hours Patients who will be operated under general anesthesia will be included.

-

Exclusion Criteria:

PATIENT DOESN'T WANT CONTRAINDICATION OF PROPOFOL Propofol allergy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: VOLUNTARY PATIENTS BETWEEN 18-65 YEARS WITH NO ADDITIONAL DISEASES
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2024-05-15 (Estimated); Primary Completion 2024-10-15 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
PROPOFOL DOSE | 2
  THE RATIO OF PROPOFOL DOSE WITH SUFFICIENT DEPTH OF ANESTHESIA ACCORDING TO TOTAL AND LEATHER BODY WEIGHT

CONTACTS AND LOCATIONS:
Locations (1):
- Inonu universitesi, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Barras M, Legg A. Drug dosing in obese adults. Aust Prescr. 2017 Oct;40(5):189-193. doi: 10.18773/austprescr.2017.053. Epub 2017 Oct 3. No abstract available. PMID 29109603
- [Background] Fujimoto M, Tanahira C, Nishi M, Yamamoto T. In non-obese patients, duration of action of rocuronium is directly correlated with body mass index. Can J Anaesth. 2013 Jun;60(6):552-6. doi: 10.1007/s12630-013-9914-x. Epub 2013 Mar 6. PMID 23463483
- See also: Drug dosing in obese adults — https://doi.org/10.1016/j.vas.2020.100131
- See also: In non-obese patients, duration of action of rocuronium is directly correlated with body mass index. — https://doi.org/10.1093/bja/aes368